CLINICAL TRIAL: NCT03740529
Title: A Phase 1/2 Study of Oral LOXO-305 in Patients With Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) or Non-Hodgkin Lymphoma (NHL)
Brief Title: A Study of Oral LOXO-305 in Patients With Previously Treated CLL/SLL or NHL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Loxo Oncology, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17539; 2018-003340-24 (EudraCT Number); J2N-OX-JZNA (Other: Eli Lilly and Company); LOXO-BTK-18001 (BRUIN) (Other: Eli Lilly and Company)
Expanded Access: NCT05172700 (Approved for marketing)
Record Dates: First submitted 2018-11-06; First posted 2018-11-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Waldenstrom Macroglobulinemia; Mantle Cell Lymphoma; Marginal Zone Lymphoma; B-cell Lymphoma; Small Lymphocytic Lymphoma
Keywords: Loxo; LOXO-305; BTK; Bruton's tyrosine kinase; CLL; SLL; NHL; Chronic Lymphocytic Leukemia; C481S; C481; Ibrutinib; Acalabrutinib; Zanubrutinib; BGB-3111; GS-4059; ONO-4059; Tirabrutinib; Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Waldenstrom macroglobulinemia; Non-Hodgkin Lymphoma; BTK Intolerant; C481S Mutation; Marginal zone lymphoma; DLBCL (Diffuse Large B-cell lymphoma); Follicular Lymphoma; PI3KD; Idelalisib; Umbralisib; BCL2; Venetoclax; Rituximab; Primary CNS Lymphoma; Richter's Transformation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular | interventions — pirtobrutinib; venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Phase I Dose Escalation (Pirtobrutinib Monotherapy) (Experimental): Dose Escalation and determination of MTD; multiple dose levels of pirtobrutinib to be evaluated
  Interventions: Drug: Pirtobrutinib
- Phase 2 (Pirtobrutinib Monotherapy) Cohort 3 (Experimental): CLL/SLL patients with no prior therapy.
  Interventions: Drug: Pirtobrutinib
- Phase 2 (Pirtobrutinib Monotherapy) Cohort 1 (Experimental): Non-blastoid MCL patients treated with a prior BTK-inhibitor containing regimen.
  Interventions: Drug: Pirtobrutinib
- Phase 2 (Pirtobrutinib Monotherapy) Cohort 4 (Experimental): CLL/SLL patients treated with prior therapy, BTK inhibitor naïve.
  Interventions: Drug: Pirtobrutinib
- Phase 2 (Pirtobrutinib Monotherapy) Cohort 2 (Experimental): CLL/SLL patients treated with 2 or more prior regimens, including a BTK inhibitor-containing regimen.
  Interventions: Drug: Pirtobrutinib
- Phase 2 (Pirtobrutinib Monotherapy) Cohort 5 (Experimental): WM patients treated with a prior BTK inhibitor-containing regimen.
  Interventions: Drug: Pirtobrutinib
- Phase 2 (Pirtobrutinib Monotherapy) Cohort 6 (Experimental): MZL patients treated with a prior BTK inhibitor-containing regimen.
  Interventions: Drug: Pirtobrutinib
- Phase 2 (Pirtobrutinib Monotherapy) Cohort 7 (Experimental): Defined as CLL/SLL or NHL not otherwise specified in Cohorts 1 through 6, inclusive of CLL/SLL, Richter's transformation, or low grade NHL with transformation, blastoid MCL, and patients with history of CNS involvement or primary CNS lymphoma. In the event the Sponsor electively closes Cohorts 2-4 prior to completion, patients with CLL/SLL who are ineligible to participate in or unable to access late phase studies of pirtobrutinib may be eligible to enroll in this cohort Diffuse large B-cell lymphoma (DLBCL) is excluded. MCL without prior BTK inhibitor treatment is excluded. Patients enrolling to Cohort 7 must have received one or more prior therapies or have no available approved therapy with demonstrated clinical benefit with the exception of untreated Richter's transformation, which is allowed.
  Interventions: Drug: Pirtobrutinib
- Phase 1b Dose Expansion (Pirtobrutinib Combination Therapy) Arm A (Experimental): Relapsed/Refractory CLL will receive the recommended Phase 2 dose of pirtobrutinib in combination with venetoclax
  Interventions: Drug: Pirtobrutinib; Drug: Venetoclax
- Phase 1b Dose Expansion (Pirtobrutinib Combination Therapy) Arm B (Experimental): Relapsed/Refractory CLL will receive the recommended Phase 2 dose of pirtobrutinib in combination with venetoclax and rituximab
  Interventions: Drug: Pirtobrutinib; Drug: Venetoclax; Drug: Rituximab
- Phase 1 Dose Expansion (Pirtobrutinib Monotherapy) (Experimental): Patients to receive the recommended Phase 2 dose of pirtobrutinib
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Oral
  Other Names: LOXO-305; LY3527727
Drug: Venetoclax — Oral
  Other Names: Venclexta, Venclyxto
  Arms: Phase 1b Dose Expansion (Pirtobrutinib Combination Therapy) Arm A; Phase 1b Dose Expansion (Pirtobrutinib Combination Therapy) Arm B
Drug: Rituximab — IV
  Other Names: Rituxan; MabThera
  Arms: Phase 1b Dose Expansion (Pirtobrutinib Combination Therapy) Arm B

SUMMARY:
This is an open-label, multi-center Phase 1/2 study of oral LOXO-305 (pirtobrutinib) in patients with CLL/SLL and NHL who have failed or are intolerant to standard of care.

DETAILED DESCRIPTION:
This study includes 3 parts: Phase 1 (pirtobrutinib monotherapy dose escalation and dose expansion), Phase 1b (pirtobrutinib combination therapy dose expansion), and Phase 2 (pirtobrutinib monotherapy dose expansion). In Phase 1, patients will be enrolled using an accelerated titration design. The starting dose of pirtobrutinib in oral tablet form is 25 mg/day (e.g., 25 mg once daily [QD]). Once the MTD and/or RP2D is identified in Phase 1 dose escalation, enrollment will continue to Phase 1 dose expansion and can commence to Phase 1b (Arms A and B). For Phase 2, patients will be enrolled to one of seven Phase 2 dose expansion cohorts depending on tumor histology and prior treatment history. Cycle length will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CLL/SLL, WM, or NHL intolerant to either ≥ 2 prior standard of care regimens given in combination or sequentially OR have received 1 prior BTK inhibitor-containing regimen when a BTK inhibitor is approved as first line therapy (Phase 1) OR with prior treatment defined by phase 2 cohort (Phase 2 Patients only).
* Adequate hematologic function (Phase 1 and 1b Patients only).
* Responsive to transfusion support if given for thrombocytopenia or anemia (Phase 1 and 1b Patients only).
* Histologically confirmed relapsed/recurrent CLL in whom venetoclax is appropriate standard salvage treatment; no prior venetoclax is permitted (Phase 1b Arm A Patients only).
* Histologically confirmed relapsed/refractory CLL in whom venetoclax + rituximab is appropriate standard salvage treatment; no prior venetoclax is permitted (Phase 1b Arm B Patients only).
* Eastern Cooperative Oncology Group (ECOG) 0-2.
* Adequate hepatic and renal function.
* Ability to receive study drug therapy orally.
* Willingness of men and women of reproductive potential (defined as following menarche and not postmenopausal [and 2 years of non-therapy-induced amenorrhea] or surgically sterile) to observe conventional and effective birth control.

Exclusion Criteria:

* Investigational agent or anticancer therapy within 5 half-lives or 14 days, whichever is shorter, prior to planned start of specified study therapy except antineoplastic and immunosuppressant monoclonal antibody treatment must be discontinued a minimum of 4 weeks prior to the first dose of pirtobrutinib. In addition, no concurrent systemic anticancer therapy is permitted.
* Major surgery within 4 weeks prior to planned start of specified study therapy.
* Radiotherapy with a limited field of radiation for palliation within 7 days of the first dose of study treatment.
* Pregnancy or lactation.
* Patients requiring therapeutic anticoagulation with warfarin.
* Any unresolved toxicities from prior therapy greater than CTCAE (version 5.0) Grade 2 or greater at the time of starting study treatment except for alopecia.
* History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified T-cell (CAR-T) therapy within the past 60 days (180 days before the PK trigger) prior to planned start of specified study therapy.
* Known central nervous system (CNS) involvement by systemic lymphoma. Patients with previous treatment for CNS involvement who are neurologically stable and without evidence of disease may be eligible and enrolled to phase 2 Cohort 7 if a compelling clinical rationale is provided by the Investigator and with documented Sponsor approval.
* Active uncontrolled auto-immune cytopenia where new therapy introduced or concomitant therapy escalated within the 4 weeks prior to study enrollment is required to maintain adequate blood counts.
* Clinically significant, uncontrolled cardiac, cardiovascular disease or history of myocardial infarction within 6 months prior to planned start of pirtobrutinib.
* Active uncontrolled systemic bacterial, viral, fungal or parasitic infection.
* Patients who have tested positive for human immunodeficiency virus (HIV) are excluded. For patients with unknown HIV status, HIV testing will be performed at Screening and result should be negative for enrollment.
* Clinically significant active malabsorption syndrome.
* Current treatment with certain strong CYP3A4 inhibitors or inducers and/or strong P-gp inhibitors.
* For patients enrolled to phase 1b Arm A or B: Patients with prior treatment with venetoclax or other BCL-2 inhibitors.
* Prior treatment with pirtobrutinib.
* Active second malignancy unless in remission and with life expectancy > 2 years.
* Known hypersensitivity to any component or excipient of pirtobrutinib.
* For patients enrolled to phase 1b Arm B: Patients with prior significant hypersensitivity, allergy, or anaphylactic reaction to rituximab/biosimilar requiring discontinuation.
* Patients with prior significant hypersensitivity to rituximab requiring discontinuation, prior allergic or anaphylactic reaction to rituximab (Phase 1b Arm B Patients only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 24 Months
  Phase I
Recommended dose for further study | Up to 24 Months
  Phase I
To assess the preliminary anti-tumor activity of pirtobrutinib based on ORR as assessed by an Independent Review Committee (IRC). | Up to 24 months
  Phase II
To evaluate the safety of pirtobrutinib in combination with venetoclax (Arm A) by assessing incidence and severity of treatment-emergent adverse events as determined by CTCAE v5.0 | Up to 24 Months
  For Phase 1b
To evaluate the safety of pirtobrutinib in combination with venetoclax and rituximab (Arm B) by assessing incidence and severity of treatment-emergent adverse events as determined by CTCAE v5.0 | Up to 24 Months
  For Phase 1b

SECONDARY OUTCOMES:
To determine the safety profile and tolerability of pirtobrutinib including acute and chronic toxicities by collecting and evaluating Adverse events and treatment emergent adverse events. | Up to 24 Months
  Phase I
To characterize the pharmacokinetics (PK) properties of pirtobrutinib by collecting and evaluating serum at protocol specified time points. | Up to 24 Months
  Phase I
To assess the preliminary anti-tumor activity of pirtobrutinib based on overall response rate (ORR) as assessed by investigator. | Up to 24 Months
  Phase I
ORR as assessed by the Investigator. | Up to 24 Months
  Phase II
Best overall response (BOR) as assessed by the Investigator and IRC. | Up to 24 Months
  Phase II
Duration of response (DOR) as assessed by the Investigator and IRC. | Up to 24 Months
  Phase II
Progression free survival (PFS) as assessed by the Investigator and IRC. | Up to 24 Months
  Phase II
Overall survival (OS). | Up to 24 Months
  Phase II
To determine the safety profile and tolerability of pirtobrutinib including acute and chronic toxicities by collecting and evaluating Adverse events and treatment emergent adverse events | Up to 24 Months
  Phase II
To characterize the pharmacokinetics (PK) properties of pirtobrutinib by collecting and evaluating serum at protocol specified time points. | Up to 24 Months
  Phase II
To characterize the pharmacokinetics (PK) properties of pirtobrutinib by collecting and evaluating serum at protocol specified time points. | Up to 24 months
  For Phase 1b
To assess the preliminary anti-tumor activity of pirtobrutinib in combination based on overall response rate (ORR) as assessed by investigator. | Up to 24 months
  For Phase 1b
Symptomatic Response: Change from Baseline in Mantle Cell Lymphoma (MCL)-related symptoms selected from the European Organisation for Research and Treatment of Cancer (EORTC) Item Library | Baseline, End of Treatment (Estimated Up to 24 Months)
  Individual EORTC symptom scores range from 1 (not at all) to 4 (very much) with higher scores representing more severe symptom severity.
Functional Response: Change from Baseline in Physical Functioning as Measured by Physical Functioning Scale from the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Version 3.0 (EORTC QLQ) | Baseline, End of Treatment (Estimated Up to 24 Months)
  EORTC physical function item scores range from 1 (not at all) to 4 (very much) with higher scores indicating poorer functioning.The total EORTC physical functioning score ranges from 0-100 where a higher score indicates higher/healthier level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Tsai, MD, PhD, Study Director — Loxo Oncology
Locations (56):
- United States (31):
  - Mayo Clinic of Scottsdale, Scottsdale, Arizona
  - Scripps Coastal Medical Center, San Diego, California
  - University of California San Francisco, Medical Center at Paranassus, San Francisco, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Florida Cancer Specialists ORLANDO/DDU, Lake Mary, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Emory Clinic, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Flinders Medical Centre, Bedford Park, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes, France
- Italy (2):
  - IRCCS - AOU di Bologna, Bologna
  - IRCCS Ospedale San Raffaele, Milan
- Japan (10):
  - Nagoya Medical Center, Nagoya, Aichi-ken
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tokai University Hospital- Isehara Campus, Isehara, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Tohoku University Hospital, Sendai, Miyagi
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyoto Furitsu Medical University Hospital, Kyoto
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Osakasayama-Shi
- Poland (2):
  - Pratia MCM Krakow, Krakow
  - Instytut Hermatologii I Transfuzjologii, Warsaw
- South Korea (2):
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Seoul National University Hospital, Seoul
- Karolinska Institutet, Solna, AB, Sweden
- Ospedale Regionale Bellinzona e Valli, Bellinzona, Canton Ticino, Switzerland
- United Kingdom (3):
  - St James's University Hospital, Leeds
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Patel K, Vose JM, Nasta SD, Brown JR, Maddocks KJ, Woyach JA, Shah NN, Fakhri B, Tessoulin B, Ma S, Jagadeesh D, Lech-Maranda E, Coombs CC, Patel MR, Rhodes JM, Ujjani CS, Hoffmann MS, Cheah CY, Munir T, Lewis DJ, Scarfo L, Eyre TA, Alencar AJ, Cohen JB, Zelenetz AD, Tsai DE, Li M, Bian Y, Abada PB, Balbas M, Zinzani PLL. Pirtobrutinib, a Highly Selective, Non-covalent (Reversible) BTKi in R/R Marginal Zone Lymphoma: Phase 1/2 BRUIN Study. Blood Adv. 2026 Jan 16:bloodadvances.2025017489. doi: 10.1182/bloodadvances.2025017489. Online ahead of print. PMID 41544219
- [Derived] Brown JR, Nguyen B, Desikan SP, Won H, Tantawy SI, McNeely SC, Marella N, Randeria HS, Hanson LM, Parker A, Botelho SC, Woyach JA, Patel K, Tam CS, Eyre TA, Cheah CY, Shah NN, Ghia P, Jurczak W, Balbas M, Nair B, Abada P, Wang C, Wang D, Roeker LE, Gandhi V, Wierda WG. Genomic determinants of response and resistance to pirtobrutinib in relapsed/refractory chronic lymphocytic leukemia. Blood. 2026 Jan 1;147(1):24-34. doi: 10.1182/blood.2024027009. PMID 41055698
- [Derived] Shah NN, Zinzani PL, Wang M, Nasta SD, Lech-Maranda E, Ogawa Y, Fakhri B, Kuss B, Miyashita K, Patel K, Coombs CC, Ma S, Patel MR, Barve MA, Tessoulin B, Stathis A, Ennishi D, Hashimoto D, Kojima K, Zelenetz AD, Cohen JB, Vose JM, Maddocks KJ, Munir T, Sun F, Bian Y, Balbas M, Tsai DE, Abada P, Cheah CY. Pirtobrutinib, a highly selective, noncovalent (reversible) BTKi in R/R follicular lymphoma: phase 1/2 BRUIN study. Blood Adv. 2025 Dec 9;9(23):5954-5964. doi: 10.1182/bloodadvances.2024014975. PMID 40845254
- [Derived] Lamanna N, Tam CS, Woyach JA, Alencar AJ, Palomba ML, Zinzani PL, Flinn IW, Fakhri B, Cohen JB, Kontos A, Konig H, Ruppert AS, Chatterjee A, Sizelove R, Compte L, Tsai DE, Jurczak W. Evaluation of bleeding risk in patients who received pirtobrutinib in the presence or absence of antithrombotic therapy. EJHaem. 2024 Sep 27;5(5):929-939. doi: 10.1002/jha2.1013. eCollection 2024 Oct. PMID 39415923
- [Derived] Wierda WG, Shah NN, Cheah CY, Lewis D, Hoffmann MS, Coombs CC, Lamanna N, Ma S, Jagadeesh D, Munir T, Wang Y, Eyre TA, Rhodes JM, McKinney M, Lech-Maranda E, Tam CS, Jurczak W, Izutsu K, Alencar AJ, Patel MR, Seymour JF, Woyach JA, Thompson PA, Abada PB, Ho C, McNeely SC, Marella N, Nguyen B, Wang C, Ruppert AS, Nair B, Liu H, Tsai DE, Roeker LE, Ghia P. Pirtobrutinib, a highly selective, non-covalent (reversible) BTK inhibitor in patients with B-cell malignancies: analysis of the Richter transformation subgroup from the multicentre, open-label, phase 1/2 BRUIN study. Lancet Haematol. 2024 Sep;11(9):e682-e692. doi: 10.1016/S2352-3026(24)00172-8. Epub 2024 Jul 18. PMID 39033770
- [Derived] Roeker LE, Woyach JA, Cheah CY, Coombs CC, Shah NN, Wierda WG, Patel MR, Lamanna N, Tsai DE, Nair B, Wang C, Zhao X, Liu D, Radtke D, Chapman S, Marella N, McNeely SC, Brown JR. Fixed-duration pirtobrutinib plus venetoclax with or without rituximab in relapsed/refractory CLL: the phase 1b BRUIN trial. Blood. 2024 Sep 26;144(13):1374-1386. doi: 10.1182/blood.2024024510. PMID 38861666
- [Derived] Telaraja D, Kasamon YL, Collazo JS, Leong R, Wang K, Li P, Dahmane E, Yang Y, Earp J, Grimstein M, Rodriguez LR, Theoret MR, Gormley NJ. FDA Approval Summary: Pirtobrutinib for Relapsed or Refractory Mantle Cell Lymphoma. Clin Cancer Res. 2024 Jan 5;30(1):17-22. doi: 10.1158/1078-0432.CCR-23-1272. PMID 37624619
- [Derived] Mato AR, Woyach JA, Brown JR, Ghia P, Patel K, Eyre TA, Munir T, Lech-Maranda E, Lamanna N, Tam CS, Shah NN, Coombs CC, Ujjani CS, Fakhri B, Cheah CY, Patel MR, Alencar AJ, Cohen JB, Gerson JN, Flinn IW, Ma S, Jagadeesh D, Rhodes JM, Hernandez-Ilizaliturri F, Zinzani PL, Seymour JF, Balbas M, Nair B, Abada P, Wang C, Ruppert AS, Wang D, Tsai DE, Wierda WG, Jurczak W. Pirtobrutinib after a Covalent BTK Inhibitor in Chronic Lymphocytic Leukemia. N Engl J Med. 2023 Jul 6;389(1):33-44. doi: 10.1056/NEJMoa2300696. PMID 37407001
- [Derived] Wang ML, Jurczak W, Zinzani PL, Eyre TA, Cheah CY, Ujjani CS, Koh Y, Izutsu K, Gerson JN, Flinn I, Tessoulin B, Alencar AJ, Ma S, Lewis D, Lech-Maranda E, Rhodes J, Patel K, Maddocks K, Lamanna N, Wang Y, Tam CS, Munir T, Nagai H, Hernandez-Ilizaliturri F, Kumar A, Fenske TS, Seymour JF, Zelenetz AD, Nair B, Tsai DE, Balbas M, Walgren RA, Abada P, Wang C, Zhao J, Mato AR, Shah NN. Pirtobrutinib in Covalent Bruton Tyrosine Kinase Inhibitor Pretreated Mantle-Cell Lymphoma. J Clin Oncol. 2023 Aug 20;41(24):3988-3997. doi: 10.1200/JCO.23.00562. Epub 2023 May 16. PMID 37192437
- [Derived] Aslan B, Kismali G, Iles LR, Manyam GC, Ayres ML, Chen LS, Gagea M, Bertilaccio MTS, Wierda WG, Gandhi V. Pirtobrutinib inhibits wild-type and mutant Bruton's tyrosine kinase-mediated signaling in chronic lymphocytic leukemia. Blood Cancer J. 2022 May 20;12(5):80. doi: 10.1038/s41408-022-00675-9. PMID 35595730
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557
- [Derived] Mato AR, Shah NN, Jurczak W, Cheah CY, Pagel JM, Woyach JA, Fakhri B, Eyre TA, Lamanna N, Patel MR, Alencar A, Lech-Maranda E, Wierda WG, Coombs CC, Gerson JN, Ghia P, Le Gouill S, Lewis DJ, Sundaram S, Cohen JB, Flinn IW, Tam CS, Barve MA, Kuss B, Taylor J, Abdel-Wahab O, Schuster SJ, Palomba ML, Lewis KL, Roeker LE, Davids MS, Tan XN, Fenske TS, Wallin J, Tsai DE, Ku NC, Zhu E, Chen J, Yin M, Nair B, Ebata K, Marella N, Brown JR, Wang M. Pirtobrutinib in relapsed or refractory B-cell malignancies (BRUIN): a phase 1/2 study. Lancet. 2021 Mar 6;397(10277):892-901. doi: 10.1016/S0140-6736(21)00224-5. PMID 33676628